CLINICAL TRIAL: NCT04944082
Title: Remdesivir Versus Remdesivir- Ivermectin Combination Therapy in Severe and Critically Ill Covid-19
Brief Title: Remdesivir- Ivermectin Combination Therapy in Severe Covid-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maiada K. Hashem, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Remdesivir-Ivermectin
Record Dates: First submitted 2021-06-23; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remdesivir only (No Intervention): (Dose 200 mg day one, 100 mg daily days 2-5), duration may extend to 10 days of remdesivir (200 mg day one, 100 mg daily days 2-10)
- Combination remdesivir plus ivermectin group (Experimental): (The same remdesivir dose as mentioned + ivermectin 4 tablet (6mg) once daily before meal for four days)
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — (The same remdesivir dose as mentioned + ivermectin 4 tablet (6mg) once daily before meal for four days)
  Arms: Combination remdesivir plus ivermectin group

SUMMARY:
Recent study reported in vitro synergistic interaction between two FDA approved drugs, remdesivir (RDV) and ivermectin (IVM) resulting in enhanced antiviral activity against SARS-CoV-2, the causative pathogen of COVID-19. The aim of the current study is comparing the efficacy and safety of combining remdesivir and ivermectin versus using remdesivir alone in patients with severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult, hospitalized severe COVID-19 patients; both genders; given informed consent (COVID-19 infection confirmed by PCR, severe illness is defined as patients with SpO2 ≤94% on room air, including patients on supplemental oxygen).

Exclusion Criteria:

* patients under 18 years old, pregnant ladies, advanced renal diseases (cr. Clearance < 30 ml/hr), raised liver enzymes> 3 folds of normal, arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
1- Improvement in level of oxygenation | By arterial blood gas and non-invasive pulse oximeter at date of randomisation, after 1 hour then on daily bases in stable cases till time of patient discharge or death
  Change in partial pressure of Oxygen and oxygen saturation
2- Need for ventilator support | From date of randomisation to patient discharge from hospital or death.
  either noninvasive or invasive mechanical ventilation.
3- Length of hospital stay | From date of randomisation to date of patient discharge from hospital or death.
  duration of admission in days
4- Development of complication | From starting to the end of ivermectin therapy (0 to the end of 4th day)
  allergic reactions, arrhythmia, hepatic toxicity.....
5- Mortality | Through study completion, an average of 3 months
  mortality rates in both groups

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Background] Pizzorno A, Padey B, Dubois J, Julien T, Traversier A, Duliere V, Brun P, Lina B, Rosa-Calatrava M, Terrier O. In vitro evaluation of antiviral activity of single and combined repurposable drugs against SARS-CoV-2. Antiviral Res. 2020 Sep;181:104878. doi: 10.1016/j.antiviral.2020.104878. Epub 2020 Jul 15. PMID 32679055